CLINICAL TRIAL: NCT01202903
Title: A 24-week, Phase III Randomized, Double-blind, Placebocontrolled, Parallel-group, Multicenter Study of Xolair® (Omalizumab) in Patients With Moderate to Severe Persistent Allergic Asthma Who Remain Not Adequately Controlled Despite GINA (2009) Step 4 Therapy
Brief Title: Omalizumab in Patients With Moderate to Severe Persistent Allergic Asthma Not Adequately Controlled Despite GINA (2009) Step 4 Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025A2313
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Persistent Allergic Asthma
Keywords: omalizumab; asthma; immunoglobulin E; IgE
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omalizumab (Experimental): Omalizumab was supplied as lyophilized, sterile powder in a single-use, 5 mL vial that was designed to deliver 150 mg of omalizumab for subcutaneous administration upon reconstitution with 1.4 mL sterile water for injection. The minimum dose of 0.016 mg/kg/IgE (IU/mL) omalizumab was administered every 4 weeks by subcutaneous injection.
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): The placebo was the same mixture of inactive excipients, in quality and quantity, as those used for the drug product. The minimum dose of 0.016 mg/kg/IgE (IU/mL) placebo was administered every 4 weeks by subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — The minimum dose of 0.016 mg/kg/IgE (IU/mL) omalizumab was administered every 4 weeks by subcutaneous injection.
  Arms: Omalizumab
Drug: Placebo — The minimum dose of 0.016 mg/kg/IgE (IU/mL) placebo was administered every 4 weeks by subcutaneous injection.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy, safety and tolerability of omalizumab, compared to placebo in 18 to 75 year old Chinese patients with moderate to severe persistent allergic asthma who have inadequate asthma control despite treatment according to GINA (2009) Step 4 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Met study drug-dosing table eligibility criteria (serum baseline total IgE level ≥ 30 to ≤ 700 IU/mL and body weight > 20 kg and ≤ 150 kg)
* Diagnosed with asthma ≥ 1 year duration at Screening, and a history of asthma that is not adequately controlled with GINA (2009) Step 4 therapy
* Received medium-to-high dose inhaled corticosteroid > 500 µg Beclomethasone Diproprionate (BDP), or equivalent plus regularly inhaled LABA, either separately or in combination, for at least 8 weeks prior to screening
* Met specific asthma exacerbations eligibility criteria prior to the screening period
* Exhibited inadequate symptom control as demonstrated by specific criteria (in keeping with GINA 2009 guidelines)
* Positive skin prick test to at least one perennial aeroallergen documented by a historical test within 12 months prior to screening, or at Visit 1
* FEV1 ≥ 40% and < 80% of the predicted normal value for the patient (using local standards), after withholding bronchodilators at Visit 2

Exclusion Criteria:

* Used other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer. For biological agent-based investigational drugs, such as monoclonal antibodies, at least six months will need to have passed between the last administration of the drug and the patient's Screening Visit.
* History of malignancy
* History of allergies and diseases that could interfere with the analyses
* Clinically significant abnormality on a 12-lead ECG recorded at Visit 1
* Elevated IgE levels for reasons other than allergy
* Current smokers, or a former smoker with a smoking history of > 10 pack-years. A former smoker must have abstained for a minimum of 12 months before randomization
* Receiving specific medications
* Clinically significant laboratory abnormalities (not associated with the study indication) at Visit 1

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- China (22):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shengyang, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai

REFERENCES:
- [Derived] Li J, Wang C, Liu C, Kang J, Kong L, Huang Y, Liu S, Huang M, Wang L, Fogel R, Jaumont X, Yang J, Zhong N. Efficacy predictors of omalizumab in Chinese patients with moderate-to-severe allergic asthma: Findings from a post-hoc analysis of a randomised phase III study. World Allergy Organ J. 2020 Nov 24;13(12):100469. doi: 10.1016/j.waojou.2020.100469. eCollection 2020 Dec. PMID 34611470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 616 patients randomized 7 (2 omalizumab and 5 placebo) did not receive drug and were excluded from the Full Analysis Set (FAS) and Safety Set.
Pre-assignment Details: One additional patient did not receive study drug for greater than 60 days and was also removed from the FAS. 4 patients initially randomized to the placebo group received omalizumab at one or more administration and were considered part of the omalizumab group for the Safety Set.
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 308 | 308
Full Analysis Set | 306 | 302
Safety Set* | 310 | 299
Completed | 297 | 292
Not Completed | 11 | 16
Not completed — Administrative Probelms | 1 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 3
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Population: The Safety Set consisted of all patients who received at least one dose of study medication whether or not being randomized. Patients were analyzed according to the treatment they actually received. If patients switched between placebo and omalizumab during the study, they were analyzed according to omalizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 310 | 299 | 609
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (12.03) | 47.1 (11.64) | 46.5 (11.85)
Age, Customized [Number; unit: Participants]
  18-<65 years | 290 | 285 | 575
  65<=75 years | 20 | 14 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 157 | 328
  Male | 139 | 142 | 281

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Morning Peak Expiratory Flow (PEF) Following the 24-week Treatment Period
Description: A Peak Expiratory Flow (PEF) meter was distributed to patients at Visit 1, to be used to measure PEF twice-daily as directed. During the Screening and Treatment Periods, PEF was measured in the morning and evening every day. the morning PEF was performed within 15 minutes after waking, and the evening PEF approximately 12 hours later. Patients were encouraged to perform morning and evening PEF measurements before the use of any LABA or rescue medication. The highest of 3 values was recorded as the daily personal best. The personal best was used to calculate the mean morning PEF and mean evening PEF value collected between assessment Visits LS Mean of change from baseline in mean morning PEF is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, gender, center grouping, smoking status, and baseline mean morning PEF as covariates.
Time Frame: Baseline, 24 weeks
Population: The FAS consisted of all randomized patients who received at least one dose of study drug. 7 randomized patients did not receive study drug and were excluded along with 1 other patient who did not receive study drug for more than 60 days
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
L/min | 27.03 (20.865) | 18.18 (21.086)

2. Secondary Outcome: Change From Baseline in Mean Evening PEF (L/Min) Following 24-week Treatment
Description: A Peak Expiratory Flow (PEF) meter was distributed to patients at Visit 1, to be used to measure PEF twice-daily as directed. During the Screening and Treatment Periods, PEF was measured in the morning and evening every day. the morning PEF was performed within 15 minutes after waking, and the evening PEF approximately 12 hours later. Patients were encouraged to perform morning and evening PEF measurements before the use of any LABA or rescue medication. The highest of 3 values was recorded as the daily personal best. The personal best was used to calculate the mean morning PEF and mean evening PEF value collected between assessment Visits. LS Mean of change from baseline in mean morning PEF is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, gender, center grouping, smoking status, and baseline mean morning PEF as covariates.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 292 | 289
L/min | 22.96 (20.145) | 15.53 (20.350)

3. Secondary Outcome: Change From Baseline in % Predicted FEV1 Following 24-week Treatment
Description: Spirometry was used at defined time points throughout the study to assess the clinical status of patients and to capture the following variables: forced expiratory volume in one second (FEV1), FEV1 percent predicted, forced vital capacity (FVC) and the FEV1/FVC ratio. During the Screening assessment, spirometry was performed pre- and post-bronchodilator administration to assess reversibility. During the treatment period (including prerandomization assessments on Day 1), spirometry was performed after withholding bronchodilators. The results of spirometry were required to meet the ATS/ERS criteria for acceptability and repeatability. Acceptability criteria were applied before repeatability was determined. LS Mean of change from baseline in % predicted FEV1 is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, gender, center grouping, smoking status, and baseline % predicted FEV1 as covariates.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
L/min | 19.113 (5.6130) | 14.989 (5.6645)

4. Secondary Outcome: Change From Baseline in AQLQ Score Following 24-week Treatment
Description: The standardized version of the Asthma Quality of Life Questionnaire (AQLQs)), was used to assess the patients' asthma-related quality of life. There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental exposure). Each question was answered on a 7 point scale (1-totally limited/problems all the time, 7-not at all limited/no problems). The overall AQLQ score is the mean of all 32 responses, and the individual domain scores are the means of the items in those domains (a minimum domain / overall score of 1 = Severely impaired whereas a maximum domain / overall score of 7 = not impaired at all). A positive change from baseline score indicates improvement.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
Units on a scale
  Overall Score (n=182,178) | 0.51 (0.155) | 0.10 (0.155)
  Symptom Score (n=208,206) | 0.47 (0.143) | 0.18 (0.142)
  Activity Score (n=203,198) | 0.46 (0.133) | 0.17 (0.131)
  Emotions Score (n=217,213) | 0.64 (0.184) | 0.36 (0.181)
  Environmental Score (n=201,203) | 0.54 (0.199) | 0.17 (0.199)

5. Secondary Outcome: Percentage of Patients Achieving at Least a 0.5, 1.0 or 1.5 Point Improvement From Baseline in AQLQ Overall Score Following 24-week Treatment
Description: as for outcome 4
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percent
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
Percent
  >=0.5 to <1.0 | 12.1 | 10.6
  >=1.0 to <1.5 | 9.2 | 6.6
  >=1.5 | 13.4 | 6.0
  Missing | 40.5 | 41.1

6. Secondary Outcome: Change From Baseline in ACQ Score Following 24-week Treatment
Description: The Asthma Control Questionnaire (ACQ) is a questionnaire consisting of 7 questions assessing symptoms, airway caliber and rescue β2-agonist use. One value representing overall asthma control on that occasion was calculated. Decrease in scores of 0.5 or higher between ACQ assessments are considered clinically meaningful. The ACQ was completed by the patient at the Investigator's site at Visit 2 (Week 1, pre-dose), Visit 6 (after completion of 16 weeks of treatment) and at the End of Study/Early Termination visit. LS Mean of change from baseline in ACQ score is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, center grouping, smoking status, and baseline ACQ score as covariates. Score 0= totally controlled, 6= extremely poorly controlled
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 210 | 211
Units on a scale | -0.51 (0.092) | -0.34 (0.091)

7. Secondary Outcome: Percentage of Patients With at Least a 0.5 or 0.75 Point Improvement in the ACQ Score at Week 24
Description: The Asthma Control Questionnaire (ACQ) is a questionnaire consisting of 7 questions assessing symptoms, airway caliber and rescue β2-agonist use. One value representing overall asthma control on that occasion was calculated. Decrease in scores of 0.5 or higher between ACQ assessments are considered clinically meaningful. The ACQ was completed by the patient at the Investigator's site at Visit 2 (Week 1, pre-dose), Visit 6 (after completion of 16 weeks of treatment) and at the End of Study/Early Termination visit. Only patients with no more than 1 item missing are included, and the missing item was imputed by interpolation
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percent
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
Percent
  <= -0.5 ACQ improvement | 34 | 24.8
  > -0.5 ACQ improvement | 34.6 | 45.0
  <= -0.75 ACQ improvement | 23.5 | 15.2
  > -0.75 ACQ improvement | 45.1 | 54.6
  Missing | 31.4 | 30.1

8. Secondary Outcome: Change From Baseline in Asthma Symptom Scores Following 24-week Treatment
Description: Total asthma symptom score was derived for each day as the total of the morning (scale 0-1), daytime (scale 0-4) and nocturnal (scale 0-4) scores with a max score of 9. The mean score across the 28 days prior to the week 24 assessment visit was used to calculate a change from baseline. Analysis of total asthma symptom score was performed using ANCOVA model and Van-Elteren test. LS Mean of change from baseline in mean asthma symptom score is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, gender, smoking status, center grouping, and baseline mean asthma symptom scores as covariates. Decrease of score on change from baseline means improvement of asthma symptom control.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
Units on a scale
  Total symptom score (n=287,282) | -1.65 (0.462) | -1.44 (0.466)
  Night-time symptom (n=292,288) | -0.67 (0.203) | -0.55 (0.205)
  Morning symptom (n=292,288) | -0.21 (0.089) | -0.20 (0.090)
  Daytime symptom (n=292,288) | -0.79 (0.246) | -0.72 (0.248)

9. Secondary Outcome: Percentage of Participants With Investigator and Patient Global Evaluation of Treatment Effectiveness (GETE) at Weeks 16 and 24
Description: The global evaluation of treatment effectiveness (GETE) is an assessment of asthma symptom control and overall response to asthma treatment. The evaluation was performed by both investigator and patient, each using the same 5 point scale. The GETE scale ranges were as follows: excellent, good, moderate, poor and worsening. A good or excellent response on the 5 point scale indicated that a patient had responded to treatment. 1=excellent 2=good 3=moderate 4=poor 5= worsening. Responder is defined as the patient who achieved an excellent or good response. Non-responder isdefined as the patient who achieved a moderate or poor or worsening response.
Time Frame: 16 and 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percent
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
Percent
  Week 16 Investigator responder | 71.9 | 52.3
  Week 16 Investigator non-responder | 25.5 | 44.4
  Week 16 Investigator missing | 2.6 | 3.3
  Week 16 Patient responder | 70.6 | 59.6
  Week 16 Patient non-responder | 26.8 | 37.1
  Week 16 Patient Missing | 2.6 | 3.3
  Week 24 Investigator responder | 70.3 | 50.7
  Week 24 Investigator non-responder | 26.5 | 45.7
  Week 24 Investigator missing | 3.3 | 3.6
  Week 24 Patient responder | 71.9 | 61.6
  Week 24 Patient non-responder | 24.8 | 34.8
  Week 24 Patient Missing | 3.3 | 3.6

10. Secondary Outcome: Change From Baseline in Number of Puffs of Asthma Rescue Medication Following 24-week Treatment
Description: Analysis of rescue medication use followed a similar method to that employed for total asthma symptom score. The mean number of puffs across the 28 days prior to the Week 24 assessment visit was used to calculate a change from baseline. LS Mean of change from baseline in mean number of puffs of asthma rescue medication is calculated with the ANCOVA model using treatment, stratification group, dosing schedule, gender, smoking status, center grouping, and baseline mean number of puffs of asthma rescue medication as covariates.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 306 | 302
Number of puffs
  Daily number of puffs (n=296,291) | -1.14 (0.566) | -0.85 (0.572)
  Daytime number of puffs (n=292-289) | -0.53 (0.301) | -0.38 (0.304)
  Nighttime number of puffs (n=292-289) | -0.56 (0.276) | -0.42 (0.279)

ADVERSE EVENTS:
Description: The Safety Set consisted of all patients who received at least one dose of study medication whether or not being randomized. Patients were analyzed according to the treatment they actually received. If patients switched between placebo and omalizumab during the study, they were analyzed according to omalizumab.
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 8/310 | 11/299
Other Adverse Events (participants affected / at risk) | 95/310 | 90/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=310) | Placebo (N=299)
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=310) | Placebo (N=299)
Pyrexia (General disorders) | 4 | 2
Influenza (Infections and infestations) | 3 | 5
Nasopharyngitis (Infections and infestations) | 20 | 26
Upper respiratory tract infection (Infections and infestations) | 40 | 38
Dizziness (Nervous system disorders) | 5 | 2
Headache (Nervous system disorders) | 3 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 31 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.